CLINICAL TRIAL: NCT05655130
Title: Effects of Peri-Operative Glucosteroid Administration on Outcomes Following Distal Radius Fracture
Brief Title: Distal Radius Steroid
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low participation rate
Sponsor: Indiana Hand to Shoulder Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R20180096
Record Dates: First submitted 2022-12-06; First posted 2022-12-19 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Fractures, Bone; Fractures, Closed; Radius Fracture Distal
MeSH Terms: conditions — Fractures, Bone; Fractures, Closed; Wrist Fractures | interventions — Dexamethasone; Methylprednisolone; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Test Group will receive 10mg intravenous dexamethasone at the time of incision, administered by the assigned anesthesiologist. Post-surgery, Test Group patients will be prescribed a 6-day oral methylprednisolone taper course.
  Interventions: Drug: Dexamethasone; Drug: Methylprednisolone
- Control Group (Other): Standard of care with no placebo
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: Dexamethasone — Intraoperative 10 mg IV Dose
  Arms: Test Group
Drug: Methylprednisolone — The oral methylprednisolone taper course will begin on the day of surgery and will taper as noted below:
  Day 1: 24 mg orally (8 mg before breakfast; 4 mg after lunch; 4 mg after dinner; 8 mg at bedtime) Day 2: 20 mg orally (4 mg before breakfast; 4 mg after lunch; 4 mg after dinner; 8 mg at bedtime) Day 3: 16 mg orally (4 mg before breakfast; 4 mg after lunch; 4 mg after dinner; 4 mg at bedtime) Day 4: 12 mg orally (4 mg before breakfast; 4 mg after lunch; 4 mg at bedtime) Day 5: 8 mg orally (4 mg before breakfast; 4 mg at bedtime) Day 6: 4 mg orally (4 mg before breakfast)
  Arms: Test Group
Other: Standard of Care — standard of care surgery
  Arms: Control Group

SUMMARY:
The primary goal of this study is to compare functional outcomes (range of motion [flexion, extension, supination, pronation], return to work, of patients with distal radius fractures who receive intraoperative glucocorticoids to those that do not. Secondary goals include comparison of pain control (number of pain pills consumed, visual analog scale (VAS) pain scores) between patients with distal radius fractures who receive intraoperative glucocorticoids to those that do not. The primary endpoint of this study will occur when 18 patients in each test-group complete the 6 month follow up visit for study.

DETAILED DESCRIPTION:
This will be a prospective, randomized, partially blinded, controlled trial where patients are randomized in a centralized fashion into 2 groups: a) Control group with no intraoperative glucocorticoids administered or b) Test group with administration of 10 mg glucocorticoids intraoperatively followed with a 6-day oral methylprednisolone taper course prescribed as a Medrol Dose Pack. Each group will enroll 30 patients for a study total of 60 over approximately a one year enrollment period. Randomization will be set up using sealedenvelope.com simple randomizer. The randomization process will ensure balance between both arms based on sex and age of patients enrolled. All patients scheduled for distal radius ORIF will be screened to meet inclusion/exclusion criteria. Patients will be randomized preoperatively by the research coordinator, based on a 1:1 weighting, upon obtaining to consent to either Control or Test group. Post-op therapists will be blinded to the patient treatment group until completion of protocol activities for each patient.

After surgery, patients will be followed for a duration of at least 6 months. Interval follow-up information will be collected at 10 days, 6 weeks, 3 months, and 6 months.

3-view wrist radiographs will be taken at each follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Intra- or extra-articular distal radius fractures (AO 23-A2,3; 23B-1,2,3; 23C-1,2,3) treated with open reduction internal fixation (ORIF)
* Age >18

Exclusion Criteria:

* Open fractures
* Pathologic fractures
* Concomitant ipsilateral upper extremity fracture (not including distal ulna)
* Medical contraindication to systemic glucocorticoids (insulin-dependent Diabetes mellitus, history of avascular necrosis, allergy)
* Narcotic dependence
* Women who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
Range of Motion | comparison of 10 days to 6 months post-operative measurements
  Active and Passive degrees of flexion, extension in the wrist. Forearm degrees of supination and pronation

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) Pain | 6 Months
  patient rates pain on a visual scale from no pain to worst possible pain

OTHER OUTCOMES:
Return to Work | 6 months
  comparison of patient's work schedule/limitations from baseline to 6 months (off study)

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana Hand to Shoulder Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No